CLINICAL TRIAL: NCT03200236
Title: Integrating Evidence-Based Smoking Cessation Interventions Into Lung Cancer Screening Programs: A Randomized Trial
Brief Title: The Lung Screening, Tobacco and Health Project
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Hackensack Meridian Health (Other); Baptist Health South Florida (Other); Lahey Hospital & Medical Center (Other); University of Michigan (Other); National Cancer Institute (NCI) (NIH); Unity Point Health (Other); MedStar Shah Medical Group (Unknown); Anne Arundel Medical Center (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016-0651; R01CA207228-01 (NIH)
Record Dates: First submitted 2017-06-19; First posted 2017-06-27 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-03

CONDITIONS: Smoking, Tobacco; Tobacco-Related Carcinoma; Tobacco Use; Lung Cancer Screening
Keywords: Lung Cancer Screening; Smoking Cessation; Tobacco Use
MeSH Terms: conditions — Tobacco Smoking; Tobacco Use; Smoking Cessation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensive Telephone Counseling (Experimental): This arm provides a multi-faceted, 8-session intensive telephone counseling (ITC) protocol, tailored on lung cancer screening results, with 8-weeks of free nicotine replacement patches provided (Nicoderm patch, 21mg, 14mg, and 7mg) and primary care engagement.
  Interventions: Behavioral: Intensive Telephone Counseling (8 sessions) with nicotine replacement
- Usual Care (Active Comparator): This arm provides a multi-faceted, 3-session usual care telephone counseling (UC) protocol, with 2-weeks of free nicotine replacement patches provided (Nicoderm patch, 21mg, 14mg, and 7mg) and primary care engagement.
  Interventions: Behavioral: Usual Care: Telephone counseling (3 sessions) with nicotine replacement

INTERVENTIONS:
Behavioral: Intensive Telephone Counseling (8 sessions) with nicotine replacement — Participants are provided up to 8 counseling sessions lasting approximately 20 minutes each and access to 8-weeks of free nicotine replacement patches. A counselor-initiated discussion of screening results will also be included throughout the counseling sessions.
  Arms: Intensive Telephone Counseling
Behavioral: Usual Care: Telephone counseling (3 sessions) with nicotine replacement — Participants are provided up to 3 counseling sessions lasting approximately 20 minutes each and access to 2-weeks of free nicotine replacement patches.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to compare intensive telephone counseling (ITC) plus the nicotine patch vs. standard telephone counseling plus the nicotine patch (Usual Care; UC) among current smokers undergoing lung cancer screening. Smoking-related outcomes will be examined at three, six and twelve months post-randomization.

DETAILED DESCRIPTION:
The investigators have built on the evidence-base of telephone counseling for smoking cessation. This pragmatic approach is designed at the intersection of scalability and intensity, for future implementation within the national tobacco quitline. In collaboration with five geographically and ethnically diverse lung cancer screening programs, the investigators will accrue smokers who have registered for screening,and are at all levels of readiness to quit. Prior to the screening day, the investigators will conduct the baseline (T0) phone interview. Following participants' receipt of their screening result (one week post-screening), the investigators will complete the T1 phone interview, provide brief advice to quit and conduct randomization. Participants will be randomized into one of two groups: ITC, in which participants are provided up to 8 counseling sessions lasting approximately 20 minutes each and access to 8-weeks of free nicotine patches. ITC will include a discussion of screening results throughout counseling sessions. The UC arm will include up to 3 counseling sessions lasting approximately 20 minutes each and access to 2-weeks of free nicotine patches. UC will not include a discussion of screening results throughout counseling sessions. All sessions will be conducted by a Tobacco Treatment Specialist (English or Spanish) and the investigators will assess intervention fidelity. In both groups, the investigators will engage referring physicians by notifying them of their patients' study enrollment and of their patients' smoking status at the 6-month follow-up. The 3-month (T2), 6-month (T3), and 12-month (T4) assessments will assess readiness to quit, quit attempts, 7-day and 30-day abstinence verified by Nicalert or carbon monoxide testing, and intervention process variables. Furthermore, two important aspects of this approach include a cost-effectiveness analysis and use of the Cancer Intervention and Surveillance Modeling Network (CISNET) to evaluate the cost of the interventions relative to their impact on short- and long-term smoking-related outcomes.

The aims are:

1. To compare ITC vs. UC standard telephone counseling. H1.1. At 3-, 6-, and 12- months, the ITC arm will have significantly improved biochemically verified 7-day and 30-day abstinence, compared to UC. H1.2. Mediators, including teachable moment factors (e.g., perceived risk based on screening results) and process measures (TC and nicotine patch adherence, primary care appointment) will positively affect cessation outcomes at 3-, 6- and 12-months. H.1.3. Moderators include screening result, readiness to quit, and nicotine dependence.
2. To evaluate reach (% of current smokers enrolled) and engagement (% who receive the interventions), both overall and among subgroups (gender, age, nicotine dependence, site). The investigators will assess intervention fidelity and feasibility for implementation, from both community-based and academically-based screening centers.
3. To conduct an economic analysis to test the hypothesis that while costlier, ITC will be more effective and have greater reach than UC in the lung screening setting, making it more cost-effective in terms of costs per 3-, 6- and 12-month cessation rates and quit attempts. The investigators will use these results as inputs to the CISNET model to project the long-term impact of the interventions on costs per life year saved and quality-adjusted life years saved, lung cancer deaths averted, lung cancer mortality reduction, and overall population mortality.

This study's strengths include the assessment of effective cessation methods designed for widespread implementation, novel components based on unique features of screening, cost-effectiveness analyses, and leveraging the University of Michigan CISNET model to project the population impact of implementing an effective cessation intervention in lung screening programs. The overall goal is to have a substantial public health impact by providing critical data to address scalability efforts by screening centers, insurers, and policy-makers.

ELIGIBILITY:
Inclusion Criteria:

* Have a >20-pack year smoking history (i.e., smoked at least a pack a day for 20 years)
* Current smokers, regardless of number smoked per day
* Can be smoking cigarettes, cigarillos, or little cigars
* English- or Spanish-speaking
* Ability to provide meaningful consent
* Have registered for CT lung cancer screening at one of our five participating lung screening sites (for enrollment) and have completed CT lung cancer screening (for subsequent follow-ups).
* Current smokers are eligible to participate regardless of prior lung cancer screening or prior cessation treatment. Smokers not yet ready to quit will be encouraged to participate.

Exclusion Criteria:

* Previously diagnosed with lung cancer
* Diagnosed with lung cancer during the study (although still eligible to receive free telephone counseling and nicotine replacement)
* At the T1 assessment when randomization occurs, individuals who have been quit for 8+ days will not be randomized. We will request that they participate in follow-up assessments of smoking status at 3-, 6- and 12-months.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1114 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Smoking cessation rate at 3-months post-randomization | Self-report measured at 3-months post-randomization; biochemical verification measured at 3-months.
  Comparison between study arms of 7-day and 30-day point prevalence cessation with biochemical verification. The investigators will also assess quit rates among subgroups (gender, age, nicotine dependence, site).
Smoking cessation rate at 6-months post-randomization | Self-report measured at 6-months post-randomization; biochemical verification measured at 6-months.
  Comparison between study arms of 7-day and 30-day point prevalence cessation with biochemical verification. The investigators will also assess quit rates among subgroups (gender, age, nicotine dependence, site).
Smoking cessation rate at 12-months post-randomization | Self-report measured at 12-months post-randomization; biochemical verification measured at 12-month assessment;
  Comparison between study arms of 7-day and 30-day point prevalence cessation. The investigators will also assess quit rates among subgroups (gender, age, nicotine dependence, site).

SECONDARY OUTCOMES:
Readiness to quit | Measured at baseline (T0), 1-2 days post-receipt of screening result (T1), and 3-months (T2), 6-months (T3), and 12-months post-randomization (T4).
  Measured using the 10-point contemplation ladder.
Quit attempts | Baseline (T0), 1-2 days post-receipt of screening result (T1),3-, 6- and 12- months post-randomization (T2, T3, T4)
  The investigators will assess the number and length of prior quit attempts at baseline. At all follow-up assessments, the investigators will assess the number and length of quit attempts that have occurred since the previous assessment.
TC intervention fidelity | Through study completion, an average of 3 months post-randomization.
  Measurement of counselor adherence to the TC protocol, which will be assessed on 10% of randomly selected participants.
Patient reach and patient engagement | Through study completion, an average of 3 months post-randomization.
  Reach: % of eligible smokers enrolled in trial; Engagement: % who receive the TC and the nicotine patch interventions), both overall and among subgroups (gender, age, nicotine dependence, site)
Costs per arm for study outcomes | Through study completion, an average of 3 months post-randomization.
  Patient time costs in the interventions; fixed costs (space, overhead) and variable costs (intervention delivery and patient participation) by arm
Cigarettes smoked per day | Measured at baseline (T0), 1-2 days post-receipt of screening result (T1), 3-months post-randomization (T2), 6 months post randomization (T3) and 12 months post randomization (T4)
  Number of cigarettes per day

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Baptist Health South Florida, Miami, Florida
  - UnityPoint Health --Trinity Medical Center, Moline, Illinois
  - Anne Arundel Medical Center, Annapolis, Maryland
  - MedStar Shah Medical Group, Hollywood, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Deidentified patient data will be shared with the National Cancer Institute as part of the SCALE collaboration.

REFERENCES:
- [Background] Taylor KL, Deros DE, Fallon S, Stephens J, Kim E, Lobo T, Davis KM, Luta G, Jayasekera J, Meza R, Stanton CA, Niaura RS, Abrams DB, McKee B, Howell J, Ramsaier M, Batlle J, Dornelas E, Parikh V, Anderson E. Study protocol for a telephone-based smoking cessation randomized controlled trial in the lung cancer screening setting: The lung screening, tobacco, and health trial. Contemp Clin Trials. 2019 Jul;82:25-35. doi: 10.1016/j.cct.2019.05.006. Epub 2019 May 23. PMID 31129371
- [Background] Cadham CJ, Cao P, Jayasekera J, Taylor KL, Levy DT, Jeon J, Elkin EB, Foley KL, Joseph A, Kong CY, Minnix JA, Rigotti NA, Toll BA, Zeliadt SB, Meza R, Mandelblatt J; CISNET-SCALE Collaboration. Cost-Effectiveness of Smoking Cessation Interventions in the Lung Cancer Screening Setting: A Simulation Study. J Natl Cancer Inst. 2021 Aug 2;113(8):1065-1073. doi: 10.1093/jnci/djab002. PMID 33484569
- [Background] Cadham CJ, Jayasekera JC, Advani SM, Fallon SJ, Stephens JL, Braithwaite D, Jeon J, Cao P, Levy DT, Meza R, Taylor KL, Mandelblatt JS; CISNET-SCALE Collaboration. Smoking cessation interventions for potential use in the lung cancer screening setting: A systematic review and meta-analysis. Lung Cancer. 2019 Sep;135:205-216. doi: 10.1016/j.lungcan.2019.06.024. Epub 2019 Jul 6. PMID 31446996
- [Result] Taylor KL, Williams RM, Li T, Luta G, Smith L, Davis KM, Stanton CA, Niaura R, Abrams D, Lobo T, Mandelblatt J, Jayasekera J, Meza R, Jeon J, Cao P, Anderson ED; Georgetown Lung Screening, Tobacco, and Health Trial. A Randomized Trial of Telephone-Based Smoking Cessation Treatment in the Lung Cancer Screening Setting. J Natl Cancer Inst. 2022 Oct 6;114(10):1410-1419. doi: 10.1093/jnci/djac127. PMID 35818122
- [Result] Cao P, Smith L, Mandelblatt JS, Jeon J, Taylor KL, Zhao A, Levy DT, Williams RM, Meza R, Jayasekera J. Cost-Effectiveness of a Telephone-Based Smoking Cessation Randomized Trial in the Lung Cancer Screening Setting. JNCI Cancer Spectr. 2022 Jul 1;6(4):pkac048. doi: 10.1093/jncics/pkac048. PMID 35818125
- [Result] Williams RM, Eyestone E, Smith L, Philips JG, Whealan J, Webster M, Li T, Luta G, Taylor KL, On Behalf Of The Lung Screening Tobacco Health Trial. Engaging Patients in Smoking Cessation Treatment within the Lung Cancer Screening Setting: Lessons Learned from an NCI SCALE Trial. Curr Oncol. 2022 Mar 23;29(4):2211-2224. doi: 10.3390/curroncol29040180. PMID 35448154
- [Result] Williams RM, Cordon M, Eyestone E, Smith L, Luta G, McKee BJ, Regis SM, Abrams DB, Niaura RS, Stanton CA, Parikh V, Taylor KL; Lung Screening, Tobacco, Health Trial. Improved motivation and readiness to quit shortly after lung cancer screening: Evidence for a teachable moment. Cancer. 2022 May 15;128(10):1976-1986. doi: 10.1002/cncr.34133. Epub 2022 Feb 10. PMID 35143041
- [Result] Eyestone E, Williams RM, Luta G, Kim E, Toll BA, Rojewski A, Neil J, Cinciripini PM, Cordon M, Foley K, Haas JS, Joseph AM, Minnix JA, Ostroff JS, Park E, Rigotti N, Sorgen L, Taylor KL. Predictors of Enrollment of Older Smokers in Six Smoking Cessation Trials in the Lung Cancer Screening Setting: The Smoking Cessation at Lung Examination (SCALE) Collaboration. Nicotine Tob Res. 2021 Nov 5;23(12):2037-2046. doi: 10.1093/ntr/ntab110. PMID 34077535
- [Result] Kim E, Williams RM, Eyestone E, Cordon M, Smith L, Davis K, Luta G, Anderson ED, McKee B, Batlle J, Ramsaier M, Howell J, Parikh V, Geronimo M, Stanton C, Niaura R, Abrams D, Taylor KL; Lung Screening, Tobacco and Health Trial. Predictors of attrition in a smoking cessation trial conducted in the lung cancer screening setting. Contemp Clin Trials. 2021 Jul;106:106429. doi: 10.1016/j.cct.2021.106429. Epub 2021 May 6. PMID 33964415
- [Result] Cordon M, Eyestone E, Hutchison S, Dunlap D, Smith L, Williams RM, Kim E, Kao JY, Hurtado-de-Mendoza A, Stanton C, Davis K, Frey J, McKee B, Parikh V, Taylor KL; Lung Screening, Tobacco, and Health Study. A qualitative study exploring older smokers' attitudes and motivation toward quitting during the COVID-19 pandemic. Prev Med Rep. 2021 Mar 11;22:101359. doi: 10.1016/j.pmedr.2021.101359. eCollection 2021 Jun. PMID 33868901